CLINICAL TRIAL: NCT04186481
Title: Safety and Performance of MINITAC◊ Ti 2.0 Suture Anchor in Extremities
Brief Title: A Study of the Safety and Performance of the MINITAC◊ Titanium 2.0 Suture Anchor
Acronym: MINITAC
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MINI.PMCF.2018.11
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Results first posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Hallux Valgus Repairs; Medial or Lateral Instability Repairs/Reconstructions; Achilles Tendon Repairs/Reconstructions; Midfoot Reconstructions; Metatarsal Ligament/Tendon Repairs/Reconstructions; Scapholunate Ligament Reconstructions; Ulnar or Radial Collateral Ligament Reconstructions; Lateral Epicondylitis Repair; Biceps Tendon Reattachment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Minitac Ti 2.0 suture anchor: Subjects who have undergone extremities repair using the Minitac Ti 2.0 Suture anchor
  Interventions: Device: MINITAC Ti 2.0 suture anchor

INTERVENTIONS:
Device: MINITAC Ti 2.0 suture anchor — The MINITAC◊ Ti 2.0 Suture Anchor is intended to provide secure reattachment of soft tissue to bone in the foot and ankle as well as elbow, wrist and hand.

SUMMARY:
This is a retrospective study evaluating the safety and performance of the MINITAC Suture anchors for extremities repair. Data will be used to support Notified Body (BSI) requirements for extremities repair indications.

DETAILED DESCRIPTION:
Up to 3 sites will participate in the study across Australia and the EU, collectively enrolling a minimum of 30 and a maximum of 50 subjects into the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has undergone extremities repair using the MINITAC◊ Ti 2.0 Suture Anchor.
2. Subject was ≥ 18 years of age at time of surgery.
3. Subject status is > 12 months post-operative.

Exclusion Criteria:

Subject is entered in another investigational drug, biologic, or device study or has been treated with an investigational product within 12 months post-operative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Thorvaldson, B.Med.Sc (Syd), B.Med.(Newc), Principal Investigator — Maitland Hand and Othopaedic surgery; Stephan Mangin, Study Chair — Clinical Director, Global Clinical Strategy, Sports Med and ENT Smith & Nephew
Locations (1):
- Maitland Hand and Othopaedic surgery, Ashtonfield, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment of this retrospective study was conducted between 25 Oct 2019 and 08 Nov 2019. 32 subjects were enrolled into the study at 1 site. All 32 subjects enrolled completed the study, of which, 31 subjects completed the 6-month visit, and 4 subjects completed the 12-month visit.
Period: Overall Study
Arm/Group | Minitac Ti 2.0 Suture Anchor
Started | 32
Completed 6 Month Visit | 31
Completed 12 Month Visit | 4
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Minitac Ti 2.0 Suture Anchor
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (14.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Black or African American | 0
  Native Hawaiian or Other Pacific Islander | 0
  White | 0
  Other | 32
  Multiple | 0
  Not Reported | 0
  Unknown | 0
Region of Enrollment [Number; unit: participants]
  Australia | 32
Height [Mean (Standard Deviation); unit: cm] | 172.19 (10.52)
Weight [Mean (Standard Deviation); unit: kg] | 83.93 (24.14)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.11 (6.42)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Success Rate (%) of the MINITAC◊ Ti 2.0 Suture Anchor in Extremities at 6 Months Post-operative
Description: Clinical success defined as extremity repairs without signs of device failure and/or reintervention as assessed by the surgeon.
Time Frame: 6 months
Population: The Full Analysis Set (FAS) included all subjects enrolled in the study who had previously undergone open or arthroscopic surgery for extremities repair using the MINITAC◊ Ti 2.0 Suture Anchor. The FAS was used for all analyses. The overall number of participants analyzed includes all participants that completed the 6 month visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Minitac Ti 2.0 Suture Anchor
Number analyzed (Participants) | 31
Participants | 31

2. Secondary Outcome: Clinical Success Rate (%) of the MINITAC◊ Ti 2.0 Suture Anchor in Extremities at 12 Months Post-operative
Description: Clinical success defined as extremity repairs without signs of device failure and/or reintervention as assessed by the surgeon for all participants that completed the 12-month visit
Time Frame: 12 months
Population: The Full Analysis Set (FAS) included all subjects enrolled in the study who had previously undergone open or arthroscopic surgery for extremities repair using the MINITAC◊ Ti 2.0 Suture Anchor. The FAS was used for all analyses. The overall number of participants analyzed includes all participants that completed the 12 month visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Minitac Ti 2.0 Suture Anchor
Number analyzed (Participants) | 4
Participants | 4

3. Other Pre Specified Outcome: Range of Motion (ROM)
Description: Range of motion defined as having full functional arc at 6 month and 12 month post-operative visits
Time Frame: 6 and 12 months
Population: The Full Analysis Set (FAS) included all subjects enrolled in the study who had previously undergone open or arthroscopic surgery for extremities repair using the MINITAC◊ Ti 2.0 Suture Anchor. The FAS was used for all analyses. The number of participants analyzed for each time frame includes all participants that completed the 6 or 12 month visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Minitac Ti 2.0 Suture Anchor
Number analyzed (Participants) | 31
Participants
  6 months - has full functional arc: Yes | 6
  6 months - has full functional arc: No | 25
  12 months - has full functional arc: number analyzed (Participants) | 4
  12 months - has full functional arc: Yes | 1
  12 months - has full functional arc: No | 3

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) and complications were collected to the extent they were available in the medical record. AE data were collected at the following timepoints: Screening - AEs from enrolment until discharge from hospital, including intraoperative complications 6 Months - AEs from discharge until 6 months follow-up 12 Months - AEs from 6 months until 12 months follow-up
Arm/Group | Minitac Ti 2.0 Suture Anchor
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 1/32
Other Adverse Events (participants affected / at risk) | 8/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minitac Ti 2.0 Suture Anchor (N=32)
Quervain's tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minitac Ti 2.0 Suture Anchor (N=32)
Bilateral MCP Joint Pain, diagnosed as Arthritis by X-ray (Musculoskeletal and connective tissue disorders) | 1 (1)
Dequervains Tensynovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Development of Small Dupuytrens Cord at level of scar over MCP joint (Musculoskeletal and connective tissue disorders) | 1 (1)
Increased Pain (General disorders) | 1 (1)
K-wire Migration (Musculoskeletal and connective tissue disorders) | 1 (1)
Lucency around Bone anchor as evidenced on X-ray (Musculoskeletal and connective tissue disorders) | 1 (1)
Mild Subluxation of Metacarpophalangeal (MCP) Joint (Musculoskeletal and connective tissue disorders) | 1 (1) — MCP Joint Mildly Subluxed With Condral Loss With The Head Of The Proximal Phalanx Rubbing Against The Head Of The Metacarpal- Left Hand
Moisture with mild Erythema to surgical wound (Musculoskeletal and connective tissue disorders) | 1 (1)
Neuropaxia around scar (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain and numbness to right thumb and radial three digits (Musculoskeletal and connective tissue disorders) | 1 (1)
Superficial infection around wire site. (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the nature of the study design, retrospective data was collected to the extent it was available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/81/NCT04186481/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT04186481/SAP_001.pdf